CLINICAL TRIAL: NCT01636726
Title: WEUKBRE5554: IMI PROTECT (Work Package 2): Use of Long Acting beta2 Adrenoceptor Agonists and Acute Myocardial Infarction (AMI)
Brief Title: WEUKBRE5554: IMI PROTECT(Work Package 2): Beta2 Agonists and Acute Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 115733; WEUKBRE5554 (Other: GSK)
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Asthma
Keywords: COPD; AMI; Asthma; LABAs
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with AMI: All patients of the study population with a record/diagnosis of AMI during the study period
  Interventions: Drug: Inhaled LABA use
- Patients without AMI: All patients of the study population without a record/diagnosis of AMI during the study period
  Interventions: Drug: Inhaled LABA use

INTERVENTIONS:
Drug: Inhaled LABA use — LABA prescription during the study period between Jan 1, 2002 and Dec 31, 2009

SUMMARY:
The studies described in this protocol are all performed within the framework of PROTECT (Pharmacoepidemiological Research on Outcomes of Therapeutics by a European ConsorTium) Work Package 2 and Workgroup 1. Primary aim of these studies is to develop, test and disseminate methodological standards for the design, conduct and analysis of Pharmacoepidemiological (PE) studies applicable to different safety issues and using different data sources. To achieve this, results from PE studies on five key adverse events (AEs) performed in different databases will be evaluated. Therefore, emphasis will be on the methodological aspects of the studies in this protocol and not on the clinical consequences of the association under investigation .

Asthma and chronic obstructive pulmonary disease (COPD) are the most common chronic airway diseases in the western world. For both, a stepwise treatment to reduce symptoms, improve lung function, and prevent risk of exacerbation is recommended using several drug classes according to guidelines published by e.g. the Global Initiative for Asthma [GINA guideline] and the Global Initiative for Chronic Obstructive Lung Disease [GOLD guideline], respectively. Beta-2-adrenoceptor agonists (B2A) are therapeutic mainstays in treating asthma and COPD due to their bronchodilative effects mediated by B2A. This drug class consists of two types of drugs: short acting B2A (SABA) which are used as a reliever medication and long acting B2A (LABA) which are used as maintenance / controller medication. Formoterol and salmeterol are the most frequently used LABA compounds with a half-life between 5-15 hrs and therefore, these compounds most commonly have labelled indications for use twice a day. .

Focussing on cardiac side effects of B2A one must consider that drugs with an opposite mechanism of action (beta-adrenoceptor-antagonists) have well-known cardio protective effects and are widely used in patients suffering from e.g. ischemic heart disease, hypertension and acute myocardial infarction (AMI)). Conversely, stimulation of cardiac beta-adrenoceptors as done by B2A may have deleterious cardiovascular effects particularly in patients with cardiac risk factors. And in fact, tachycardia and arrhythmias are well-known side effects of B2A confirming a cardiac influence of these drugs particularly after oral therapy (due to a high systemic exposure) as stated in the respective summary of product characteristics (SPCs), e.g. clenbuterol (Spiropent(R)). Obviously, inhaled drugs cause much smaller systemic exposure but cardiac side effects (e.g. arrhythmias, tachycardia) are also described in the respective SPCs (e.g. formoterol [Foradil(R)). Furthermore, cardiac side were also reported after exposure with inhaled MA (e.g. ipratropium [Atrovent(R)].

Several observational studies have been performed on the association between the usage of inhaled B2A and the occurrence of AMI. However, these studies have produced conflicting results. Reasons for this variation are numerous, e.g. small number of events (AMI) leading to poor precision of risk estimate, potential misclassification of potential cardiac events versus airway-related events due to similar clinical complaints, differences in populations of drug users, measurement of drug exposure, and background risk of AMI. Additionally, a consensus document was released in 2000, redefining AMI.

To make comparing results possible, this protocol gives guidelines for conducting studies in the same way in five databases and across 3 designs (cohort, nested case-control, case-cross-over) on the association between inhaled LABA use and AMI. The main focus is to evaluate the impact of study design, population and database characteristics on the association between inhaled LABA and AMI.

Data will be collected from the following databases: The Health Improvement Network (THIN), the General Practice Research Database (GPRD), the Dutch Mondriaan project, Base de Datos para la Investigación Farmacoepidemiológica en Atencion Primaria (BIFAP), the National Databases of Denmark, and the Bavarian statutory health insurance physicians' association database.

ELIGIBILITY:
Inclusion Criteria:

For the descriptive sudy:

* patients who have at least one documented and valid data record in the period from Jan 1, 2002 to Dec 31, 2009
* patients who have a diagnosis of asthma and/or COPD

For the cohort and nested case-control studies:

* patients who have at least one documented and valid data record in the period from Jan 1, 2002 to Dec 31, 2009
* patients who have a diagnosis of asthma and/or COPD
* patients who have at least one prescription of LABA/LAMA/SABA/SAMA

Exclusion criteria:

For the cohort and nested case-control studies:

* patients who had AMI within 1 year before the index date

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Descriptive study - all patients included in the period of valid data collection. The study period will be defined from Jan 1, 2002 to Dec 31, 2009.
  Cohort and nested case-control studies - all patients who received at least one prescription of an inhaled LABA, SABA, LAMA, or SAMA and with coded diagnosis of asthma and / or COPD during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2012-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
The first Acute Myocardial Infarction (AMI) in the study period | Up to eight years following drug exposure

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline